CLINICAL TRIAL: NCT03167424
Title: Observational Study of Treatment of Bioresorbable Vascular Scaffolds Restenosis
Brief Title: Restenosis Intrastent: Treatment of Bioresorbable Vascular Scaffolds Restenosis
Acronym: RIBS VII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Instituto de Investigación Sanitaria Hospital Universitario de la Princesa (Other); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Fernando Alfonso, MD, Principal Investigator, Spanish Society of Cardiology
Other Study IDs: RIBS VII
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Coronary In-stnent Restenosis
Keywords: In-stent restenosis; Bioresorbable vascular scaffold; Coronary angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BVS restenosis: Patients with a Bioresorbable Vascular Scaffold Restenosis
  Interventions: Device: Treatment of restenosis

INTERVENTIONS:
Device: Treatment of restenosis — Treatment of in-stent restenosis

SUMMARY:
The treatment of patients with intra-stent restenosis (ISR) of Bioresorbable Vascular Scaffolds (Abbott Vascular) remains a challenge. This study will assess the incidence, predisposing factors, pathophysiology and prognosis of the patient in this setting.

DETAILED DESCRIPTION:
Treatment of patients with ISR remains a challenge. Currently both drug-eluting stents (DES) and drug-coated balloons (DCB) are considered as the strategies of choice in this setting. However, existing data about ISR of BVS are scarce (isolated cases and retrospective series with very few patients) on the incidence, predisposing factors, pathophysiology, treatment, and long-term prognosis of these patients. In this sense, a prospective Spanish registry of patients with ISR of DVB can obtain a very relevant clinical information that allows us to advance in our knowledge about this phenomenon that helps to prevent it and to treat it in the safest and most effective way possible.

Clinical events will be adjudicated by an independent Clinical Event Committee.

ELIGIBILITY:
In-stent restenosis of BVS with ischemia. Signed Informed Consent IRB approval.

INCLUSION CRITERIA:

PATIENT

* Age > 20 and < 85 years of age
* Angina or objective evidence of ischemia LESION
* ISR (>50% diameter stenosis on visual assessment)
* Previous stent location known

EXCLUSION CRITERIA:

PATIENT

* Inclusion in other clinical research protocol
* Refuse to sign Informed Consent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-stent restenosis of bioresorbable vascular scaffold.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Combined clinical end-point (cardiac death, myocardial infarction and target vessel revascularization) | 1 year of clinical follow-yp
  This is a well-accepted outcome measure of individual clinical end-points. Definition of myocardial infarction is similar to that used in previous RIBS studies. The occurrence of ANY of these events will qualify for the combined event. That is, Cardiac death OR Myocardial Infarctio OR target vessel revascularization. (for the cobined end point the first event will be censored for each patient and other subsequent events will not apply). For time related statistics, the first event will be censored in the KM curves. In addition to that, the time and occurrence of each individual event will be also analyzed.
  The same strategy will be followed for the other combined clinical outcome measures that, again, are classically defined in this field.

SECONDARY OUTCOMES:
Target-lesion failure (defined as cardiac death, target-vessel myocardial infarction, or ischemia-driven target-lesion revascularization) | 1 year, 2 years, 3 years, 4 years, 5 years
  This is a well-accepted outcome measure of individual clinical end-points
Combined clinical outcome measure (cardiac death, myocardial infarction, target lesion revascularization) | 1 year, 2 years, 3 years, 4 years, 5 years
  This is a well-accepted outcome measure of individual clinical end-points. Definition of myocardial infarction is similar to that used in previous RIBS studies. The occurrence of ANY of these events will qualify for the combined event. That is, Cardiac death OR Myocardial Infarctio OR target vessel revascularization. (for the cobined end point the first event will be censored for each patient and other subsequent events will not apply). For time related statistics, the first event will be censored in the KM curves. In addition to that, the time and occurrence of each individual event will be also analyzed. The same strategy will be followed for the other combined clinical outcome measures that, again, are classically defined in this field.
Cardiac death | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Total mortality | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Myocardial infarction | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Target vessel revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Target lesion revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Stent thrombosis | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Major bleeding | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Complexo Universitario Hospitalario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Result] Alfonso F, Zueco J, Cequier A, Mantilla R, Bethencourt A, Lopez-Minguez JR, Angel J, Auge JM, Gomez-Recio M, Moris C, Seabra-Gomes R, Perez-Vizcayno MJ, Macaya C; Restenosis Intra-stent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. A randomized comparison of repeat stenting with balloon angioplasty in patients with in-stent restenosis. J Am Coll Cardiol. 2003 Sep 3;42(5):796-805. doi: 10.1016/s0735-1097(03)00852-0. PMID 12957423
- [Result] Alfonso F, Melgares R, Mainar V, Lezaun R, Vazquez N, Tascon J, Pomar F, Cequier A, Angel J, Perez-Vizcayno MJ, Sabate M, Banuelos C, Fernandez C, Garcia JM; Restensois Intra-stent: Ballon angioplasty versus elective Stenting (RIBS) Investigators. Therapeutic implications of in-stent restenosis located at the stent edge. Insights from the restenosis intra-stent balloon angioplasty versus elective stenting (RIBS) randomized trial. Eur Heart J. 2004 Oct;25(20):1829-35. doi: 10.1016/j.ehj.2004.07.019. PMID 15474698
- [Result] Alfonso F, Auge JM, Zueco J, Bethencourt A, Lopez-Minguez JR, Hernandez JM, Bullones JA, Calvo I, Esplugas E, Perez-Vizcayno MJ, Moreno R, Fernandez C, Hernandez R, Gama-Ribeiro V; RIBS Investigators. Long-term results (three to five years) of the Restenosis Intrastent: Balloon angioplasty versus elective Stenting (RIBS) randomized study. J Am Coll Cardiol. 2005 Sep 6;46(5):756-60. doi: 10.1016/j.jacc.2005.05.050. PMID 16139121
- [Result] Alfonso F, Perez-Vizcayno MJ, Gomez-Recio M, Insa L, Calvo I, Hernandez JM, Bullones JA, Hernandez R, Escaned J, Macaya C, Gama-Ribeiro V, Leitao-Marques A; Restenosis Intrastent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. Implications of the "watermelon seeding" phenomenon during coronary interventions for in-stent restenosis. Catheter Cardiovasc Interv. 2005 Dec;66(4):521-7. doi: 10.1002/ccd.20524. PMID 16261546
- [Result] Alfonso F, Cequier A, Angel J, Marti V, Zueco J, Bethencourt A, Mantilla R, Lopez-Minguez JR, Gomez-Recio M, Moris C, Perez-Vizcayno MJ, Fernandez C, Macaya C, Seabra-Gomes R; Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) Investigators. Value of the American College of Cardiology/American Heart Association angiographic classification of coronary lesion morphology in patients with in-stent restenosis. Insights from the Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) randomized trial. Am Heart J. 2006 Mar;151(3):681.e1-681.e9. doi: 10.1016/j.ahj.2005.10.014. PMID 16504631
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Mantilla R, Moris C, Cequier A, Sabate M, Escaned J, Moreno R, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. A randomized comparison of sirolimus-eluting stent with balloon angioplasty in patients with in-stent restenosis: results of the Restenosis Intrastent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) trial. J Am Coll Cardiol. 2006 Jun 6;47(11):2152-60. doi: 10.1016/j.jacc.2005.10.078. PMID 16750678
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Fernandez C, Escaned J, Banuelos C, Bethencourt A, Lopez-Minguez JR, Angel J, Cequier A, Sabate M, Moris C, Zueco J, Seabra-Gomes R; Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Stent Implantation (RIBS-I) and Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) Investigators. Sirolimus-eluting stents versus bare-metal stents in patients with in-stent restenosis: results of a pooled analysis of two randomized studies. Catheter Cardiovasc Interv. 2008 Oct 1;72(4):459-67. doi: 10.1002/ccd.21694. PMID 18814274
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Iniguez A, Moris C, Cequier A, Sabate M, Escaned J, Jimenez-Quevedo P, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. Long-term clinical benefit of sirolimus-eluting stents in patients with in-stent restenosis results of the RIBS-II (Restenosis Intra-stent: Balloon angioplasty vs. elective sirolimus-eluting Stenting) study. J Am Coll Cardiol. 2008 Nov 11;52(20):1621-7. doi: 10.1016/j.jacc.2008.08.025. PMID 18992651
- [Result] Alfonso F, Perez-Vizcayno MJ, Dutary J, Zueco J, Cequier A, Garcia-Touchard A, Marti V, Lozano I, Angel J, Hernandez JM, Lopez-Minguez JR, Melgares R, Moreno R, Seidelberger B, Fernandez C, Hernandez R; RIBS-III Study Investigators (under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology). Implantation of a drug-eluting stent with a different drug (switch strategy) in patients with drug-eluting stent restenosis. Results from a prospective multicenter study (RIBS III [Restenosis Intra-Stent: Balloon Angioplasty Versus Drug-Eluting Stent]). JACC Cardiovasc Interv. 2012 Jul;5(7):728-37. doi: 10.1016/j.jcin.2012.03.017. PMID 22814777
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Seidelberger B, Iniguez A, Gomez-Recio M, Masotti M, Velazquez MT, Sanchis J, Garcia-Touchard A, Zueco J, Bethencourt A, Melgares R, Cequier A, Dominguez A, Mainar V, Lopez-Minguez JR, Moreu J, Marti V, Moreno R, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS V Study Investigators, under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology. A randomized comparison of drug-eluting balloon versus everolimus-eluting stent in patients with bare-metal stent-in-stent restenosis: the RIBS V Clinical Trial (Restenosis Intra-stent of Bare Metal Stents: paclitaxel-eluting balloon vs. everolimus-eluting stent). J Am Coll Cardiol. 2014 Apr 15;63(14):1378-86. doi: 10.1016/j.jacc.2013.12.006. Epub 2014 Jan 8. PMID 24412457
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Rivero F, Masotti M, Zueco J, Cequier A, Moris C, Fernandez-Ortiz A, Escaned J, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; Restenosis Intra-stent: drug-eluting Balloon vs. everolimus-eluting Stent (RIBS IV) Study Investigators (under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology). Rationale and design of the RIBS IV randomised clinical trial (drug-eluting balloons versus everolimus-eluting stents for patients with drug-eluting stent restenosis). EuroIntervention. 2015 Jul;11(3):336-42. doi: 10.4244/EIJY14M09_07. PMID 25244700
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Benedicto A, Masotti M, Zueco J, Iniguez A, Velazquez M, Moreno R, Mainar V, Dominguez A, Pomar F, Melgares R, Rivero F, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS IV Study Investigators (under auspices of Interventional Cardiology Working Group of Spanish Society of Cardiology). A Prospective Randomized Trial of Drug-Eluting Balloons Versus Everolimus-Eluting Stents in Patients With In-Stent Restenosis of Drug-Eluting Stents: The RIBS IV Randomized Clinical Trial. J Am Coll Cardiol. 2015 Jul 7;66(1):23-33. doi: 10.1016/j.jacc.2015.04.063. PMID 26139054
- [Derived] Alfonso F, Cuesta J, Ojeda S, Camacho-Freire S, Garcia Del Blanco B, Vaquerizo B, Zueco J, Trillo R, Mauri J, Velazquez M, Cordoba-Soriano JG, Serra A, Navarro F, Pan M, Diaz J, Otaegui I, Salvatella N, De la TorreHernandez JM, Val DD, Bastante T, Rivero F; Under the auspices of the Association of Interventional Cardiology of the Spanish Society of Cardiology. Procedural Results and One-Year Clinical Outcomes of Treatment of Bioresorbable Vascular Scaffolds Restenosis (from the RIBS VII Prospective Study). Am J Cardiol. 2022 Jan 1;162:31-40. doi: 10.1016/j.amjcard.2021.09.027. PMID 34903344